CLINICAL TRIAL: NCT06494150
Title: Phase II Study of Nab-sirolimus and Endocrine Therapy in Recurrent Low Grade Serous Ovarian Cancer
Brief Title: Nab-Sirolimus and Endocrine Therapy in Recurrent Low Grade Serous Ovarian Cancer (NARETO)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-NARETO
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Low Grade Ovarian Serous Adenocarcinoma
Keywords: Ovarian Cancer; Endocrine Therapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Intervention Model Description: A single arm phase II study proposes to evaluate the efficacy and safety of nab-sirolimus + endocrine therapy in patients with recurrent LGSOC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nab-sirolimus + Fulvestrant (Experimental): Patients will be treated with the combination nab-sirolimus (100 mg/m2 intravenous injection on day 1 and 8 of each 21-day cycle) and fulvestrant (500mg intramuscular injection on days 1 and 15 of cycle 1 and then every 21 days).
  Interventions: Drug: nab-Sirolimus; Drug: Fulvestrant

INTERVENTIONS:
Drug: nab-Sirolimus — nab-Sirolimus will be administered by intravenous infusion at 100mg/m2 on days 1 and 8 of each 21-day cycle
  Other Names: Fyarro
Drug: Fulvestrant — Fulvestrant will be administered by intramuscular injection at 500mg on days 1 and 15 of cycle 1 and then every 21 days
  Other Names: Faslodex

SUMMARY:
This single arm phase II study proposes to evaluate the efficacy and safety of nab-sirolimus + endocrine therapy (Fulvestrant) in patients with recurrent low grade serous ovarian cancer (LGSOC).

DETAILED DESCRIPTION:
Patients with histologic confirmed Low Grade Serous Ovarian Cancer with measurable disease should have a pre-dose tumor biopsy.

Patients will receive proposed treatment regimen of nab-sirolimus on days 1 and 8 and fulvestrant on days 1 and 15 of cycle 1 and then every 21-day cycle as long as there is evidence that tumor is not growing or spreading and they are not having any unacceptable, bad side effects.

Patients will be monitored during treatment with tests and exams and after treatment completion for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologic confirmed low-grade serous ovarian cancer with clinical evidence of reoccurrence.
2. All patients must have measurable disease as defined by RECIST version 1.1.
3. ECOG Performance status must be 0-1.
4. Adequate bone marrow, hepatic and renal function as defined by the protocol.
5. At least 4 weeks must have elapsed since the patient underwent any major surgery.
6. At least 2 weeks must have elapsed since the patient received any radiation therapy.
7. Patients must have signed an IRN approved informed consent and authorization permitting release of personal health information.
8. All patients must be at least 18 years of age.
9. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
10. Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing a highly effective form of contraception. During the study treatment and for 12 weeks after stopping nab-sirolimus and 12 months after stopping Fulvestrant. Highly effective contraceptive methods include combination of any two of the following as defined in the protocol.

Exclusion Criteria:

1. Patients who have previously received nab-sirolimus, any other mTOR inhibitor or any agent targeting the PI3K/AKT/mTOR pathway. (Prior MEKi is not exclusionary; up to one prior cytotoxic therapy is permissible.)
2. Known intolerance or hypersensitivity to nab-sirolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus).
3. Patients receiving chronic treatment with systemic steroids or another immunosuppressive agent if >10 mg prednisone equivalent per day
4. Patients with active or uncontrolled systemic infection requiring IV antibiotics, either ongoing or completed ≤7 days prior to enrollment.
5. Known severely impaired lung function, including:

   * CTCAE grade 2 (or greater) hypoxia (decreased oxygen saturation with exercise [e.g., pulse oximeter <88%]; intermittent supplemental oxygen)
6. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification 1. To be eligible for this trial, patients should be class 2B or better.
7. Cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) within 6 months prior to the first date of study therapy.
8. Patients who are hypersensitive to albumin.
9. Patients who are pregnant or breast-feeding.
10. Patients with brain metastases. Patients recently treated for brain metastases are eligible as long as they have been off steroids or RT for at least 2 weeks.
11. Known HIV-infected patients requiring anti-retroviral therapy that are strong CYP3A4 inhibitors or inducers.
12. Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder or coagulopathy.
13. Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 28 days prior to dosing or 5 half-lives whichever is shorter.
14. Active Hepatitis B or Hepatitis C, with detectable viral load.

    * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
15. Uncontrolled hypertension (systolic blood pressure ≥160 mm-Hg and/or diastolic blood pressure ≥100 mm Hg).
16. Patients who are unable to discontinue concomitant medication with CYP3A4 strong inducers (eg, rifampin, rifabutin), and known CYP3A4 substrates with a narrow therapeutic window (eg, fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, or terfenadine) at least 5 half-lives prior to receiving the first dose of nab-sirolimus. Medical Monitor approval required if patient is taking any of the medications listed above.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
The percentage of people in a treatment group who have a partial or complete response to the treatment within a certain period of time as measured by RECIST version 1.1. | 3 years
  The primary analysis is preplanned to occur when the last patient enrolled has been treated for 6 months.
Incidence of patients with ≥ grade 3 adverse events. | 3 years
  Review of adverse events that have occurred to determine the toxicity for the proposed treatment regimen.

SECONDARY OUTCOMES:
Proportion of patients who have remained progression-free for 6-months. | 3 years
  Proportion of patients on the proposed treatment combination who have not had any disease progression for at least 6 months.
Duration of response from a subjects first scan to disease progression or death. | Up to 3 years
  Determine the length of time from the date subjects have partial or complete response to treatment until the date the subjects have disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Washington, MD, Principal Investigator — OU Health Stephenson Cancer Center
Locations (1):
- OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No